CLINICAL TRIAL: NCT00435890
Title: Randomized Controlled Trial of a Liaison Physician at the Triage Desk to Reduce Emergency Department Overcrowding and Improve Patient Flow.
Brief Title: Triage Liaison Physician - Evaluation of a Novel Approach to Address Emergency Department Overcrowding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Brian Holroyd, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B-091105
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Acute Illness
Keywords: ED Overcrowding; Length of stay; Emergency triage; triage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention): No triage liaison physician
  Interventions: Behavioral: Triage Liaison Physician

INTERVENTIONS:
Behavioral: Triage Liaison Physician — triage liaison physician stationed with nurses at the triage desk of the Emergency Department.

SUMMARY:
This randomized controlled trial will introduce a triage liaison physician (TLP) into the University of Alberta Hospital Emergency Department (ED) and assess the influence on patients who leave without being seen, ED length of stay, and other ED Overcrowding outcomes.

DETAILED DESCRIPTION:
ED Overcrowding is a significant cause of delayed care, patient dissatisfaction, and poor outcomes in North American EDs. This intervention has not been widely studied; however, it represents an opportunity for improving patient flows in EDs.

ELIGIBILITY:
Inclusion Criteria:

* Only adult patients (> 17 years of age) presenting to the University of Alberta Hospital Emergency Department (UAH ED), during the study interval will be included in the evaluation.

Exclusion Criteria:

* Direct admits/Pediatric patients.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5718 (Actual)
Dates: Start 2005-12; Primary Completion 2006-02 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Median patient length of stay | while in the Emergency Department

SECONDARY OUTCOMES:
Left without being seen | while in the Emergency Department
ambulance turnaround times | while in the Emergency Department
satisfaction (physicians and nurses) | following their Emergency Department shift
TLP activity | while in the Emergency Department

CONTACTS AND LOCATIONS:
Overall Officials: Brian H Rowe, MD, Study Director — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Holroyd BR, Bullard MJ, Latoszek K, Gordon D, Allen S, Tam S, Blitz S, Yoon P, Rowe BH. Impact of a triage liaison physician on emergency department overcrowding and throughput: a randomized controlled trial. Acad Emerg Med. 2007 Aug;14(8):702-8. doi: 10.1197/j.aem.2007.04.018. PMID 17656607